CLINICAL TRIAL: NCT01700920
Title: PHASE II CLINICAL TRIAL Prospective, Open, Nonrandomized Treatment of Osteonecrosis of the Femoral Head by the Administration of Autologous Mesenchymal Stem Cells
Acronym: CSM/ON/2011
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Red de Terapia Celular (Industry)
Collaborators: Haematology Service,University Hospital of Salamanca, MªConsuelo del Cañizo Fernández-Roldán (Other); Spanish National Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSM/ON/2011
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Osteonecrosis of the Femoral Head
Keywords: Osteonecrosis of the femoral head; Stem Cell; Mesenchymal Stem Cells; Femoral Head
MeSH Terms: conditions — Legg-Calve-Perthes Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesenchymal Stem Cell (Experimental): Cell suspension mesenchymal stem cells (MSCs) obtained from bone marrow aspirate from the patient and expanded in vitro in a specific medium enriched with platelet lysate without addition of animal products.
  They employ a minimum dose of 0.5 x 106 MSC / kg and a maximum of 1, 0x106 CSM / kg of patient weight.
  Pharmaceutical form: Suspension cell Route of administration: local implant intraosseous injection with trocar in the femoral head.
  Interventions: Procedure: bone marrow aspirate

INTERVENTIONS:
Procedure: bone marrow aspirate

SUMMARY:
The purpose of this study is to analyze the safety and feasibility of direct administration intrafemoral mesenchymal stem cells (MSCs) in vitro expanded autologous treatment of patients with femoral osteonecrosis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Clinical diagnosis and imaging (Rx and NMR) of idiopathic osteonecrosis of the femoral head
* Stadiums <IIIC ARCO ranking

Exclusion Criteria:

* Those on investigator judgment not in a good position to tolerate the procedure.
* Clinical criteria and anesthetics that contraindicate surgery (eg ASA IV-V)
* Serious illness uncontrolled
* Pregnant women
* Patients with HIV infection +
* Acute infection (in the previous 15 days) or chronic (other than HIV)
* Previous treatments of osteonecrosis
* Active or previous neoplastic disease (last 5 years) except for patients undergoing allogeneic haematopoietic progenitors who are in complete remission after 2 years after transplantation.
* Lack of informed consent or revocation thereof.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Salamanca, Salamanca, Castille and León, Spain

REFERENCES:
- See also: Spanish cell therapy network (TerCel) — http://www.red-tercel.com
- See also: Salamanca University Foundation — http://fundacion.usal.es
- See also: Spanish Health Institute Carlos III — http://www.isciii.es